CLINICAL TRIAL: NCT00547781
Title: Implantation Failure and PGD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Dr. Carmen Rubio, IVI Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VLC-JD-0704-307-12
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: IMPLANTATION
MeSH Terms: interventions — Prostaglandins D

INTERVENTIONS:
Procedure: PGD

SUMMARY:
The aim of this study is to performed a randomized controlled trial to evaluate the usefulness of preimplantation genetic diagnosis (PGD) in patients with repetitive implantation failure. Patients will be prospectively randomized in two groups: standard IVF with blastocyst transfer on day-5 and transfer day-5 after PGD for aneuploidy screening for chromosomes 13, 15, 16, 18, 21, 22, X and Y. The end points of the study are: Cancellation rate; implantation rate and ongoing implantation rate. Inclusion criteria are: patients with ≥2 previous IVF failure without clinical or biochemical pregnancy with transfer of at least 2 good quality embryos per transfer. Exclusion criteria will be uterine abnormalities , abnormal karyotypes, abnormal result in thrombophilia screening and low responder patients (less than 4 expected oocytes).

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age with ≥2 previous cycles, negative TIG or biochemical pregnancy with fresh transfer of at least 2 embryos in each cycle.

Exclusion Criteria:

* Patients with PGD indication (age, repetitive miscarriage, chromosomal anomalies, etc. )
* Patients with ectopic pregnancies in previous cycles.
* Recipient of oocyte donation.
* Patients in which 4 or less oocytes are to be retrieved.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2007-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Rubio, PhD, Principal Investigator — IVI Valencia
Locations (1):
- IVI Valencia, Valencia, Valencia, Spain